CLINICAL TRIAL: NCT03514667
Title: The Effects of Nanomicielle Curcumin on Oxidative Stress, Systemic Inflammation, Adiponectin in Serum and NF-kB in Blood Mononuclear Cells, in Patients With Metabolic Syndrome
Brief Title: The Effects of Nanocurcumin on Serum Oxidative Stress,Inflammation,Adiponectin and NF-kB in Blood Mononuclear Cells in Metabolic Syndrome Patients (Nuclear Factor-κB)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, clinical professor, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 188
Record Dates: First submitted 2018-04-20; First posted 2018-05-02 (Actual); Last update posted 2018-07-31 (Actual); Status verified 2018-07

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): 80 mg nanomicielle curcumin capsules once a day for 12 weeks
  Interventions: Dietary Supplement: nanomicielle curcumin
- control group (Placebo Comparator): placebo capsules once a day for 12 weeks
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: nanomicielle curcumin — Participants will be selected from those referring to endocrinology clinics of Shohadaye YaftAbad and Pars Hospital (Tehran, Iran) who meet the inclusion criteria. Each subject will give informed written consent to participate in the study. 10 cc fasting blood samples will be collected from each subject at baseline and at the end of trial. Anthropometric parameters will be measured.In order to control the confounding factors in patients, they will be randomly assigned to receive either nanomicielle curcumin or placebo. nanomicielle curcumin and placebo supplements will be provided from the Elixir Nano Sina Company the patients will advise not to change their lifestyle during the study.
  Arms: intervention group
Dietary Supplement: placebo — Participants will be selected from those referring to endocrinology clinics of Shohadaye YaftAbad and Pars Hospital (Tehran, Iran) who meet the inclusion criteria. Each subject will give informed written consent to participate in the study. 10 cc fasting blood samples will be collected from each subject at baseline and at the end of trial. Anthropometric parameters will be measured.In order to control the confounding factors in patients, they will be randomly assigned to receive either nanomicielle curcumin or placebo. nanomicielle curcumin and placebo supplements will be provided from the Elixir Nano Sina Company the patients will advise not to change their lifestyle during the study.
  Arms: control group

SUMMARY:
Metabolic syndrome is a public health challenge that includes a range of conditions including abdominal obesity, dyslipidemia, hyperglycemia, and hypertension. The syndrome is associated with an increase in the risk of Cardiovascular disease and death. Curcumin is a very active compound obtained from turmeric root. Curcumin has antioxidant and anti-inflammatory effects, and is also involved in the regulation of several signaling pathways. Since curcumin powder has low bioavailability, fast metabolism and low absorption, nanomicielle curcumin will be used in this study. Therefore, this study is planned to determine the effects of supplementation of nanomicielle curcumin on oxidative stress, systemic inflammation, adiponectin in serum and NF-kB in peripheral blood mononuclear cells in patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* 25<body mass index >40
* waist circumference >102 cm in men or >88 cm in women
* Fasting blood glucose >100 mg/dL
* Triglycerides (TG) > 150 mg/dL
* High density lipoprotein cholesterol (HDL-C) <50 in women or <40 in men
* Systolic blood pressure (SBP) >130 mmHg and diastolic blood pressure (DBP) >85mmHg

Exclusion Criteria:

* insulin administration for diabetes control
* hypo- or hyperthyroidism,
* renal failure or other chronic diseases
* pregnancy and breastfeeding
* taking weight loss supplements and obeying unusual weight loss plans

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-08-30 (Estimated); Primary Completion 2019-08-30 (Estimated); Study Completion 2020-01-30 (Estimated)

PRIMARY OUTCOMES:
Serum Total antioxidant capacity (TAC) | 12 weeks
Serum Malondialdehyde (MDA) | 12weeks
Serum C-reactive protein (CRP) | 12weeks
Serum Adiponectin | 12weeks
NF-kB(p65) transcription in PBMC | 12weeks
Serum curcumin | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Golbon Sohrab, Tehran, National Nutrition and Food Technology Research Institute, Iran